CLINICAL TRIAL: NCT01037595
Title: Effect of Turmeric on Pruritus in Hemodialysis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maryam Pakfetrat, associated professor of shiraz Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3441
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: End Stage Renal Failure
Keywords: hemodialysis; turmeric; pruritus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- turmeric (Experimental): turmeric 500 mg tid orally for 8 weeks
  Interventions: Drug: turmeric
- plasebo (Placebo Comparator): placebo tid orally for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: turmeric — turmeric 500 md tid orally for 8 weeks
  Arms: turmeric
Drug: placebo — placebo 3 time orally for 8 weeks
  Arms: plasebo
Drug: turmeric — 500 mg tid orally for 8 weeks
  Arms: turmeric

SUMMARY:
The purpose of this study is to see whether turmeric can be effective in treatment of pruritus in hemodialysis patients.

DETAILED DESCRIPTION:
pruritus is a common in hemodialysis patients and many treatment recommended for it . as turmeric has anti-inflammatory , anti-cytokine and anti-oxidant effect it may effective in treatment of uremic pruritus. thus we compared turmeric with placebo in this study

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis for more than 3 months
* More than 18 years old
* Pruritus

Exclusion Criteria:

* Use other treatment for pruritus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
improvement in pruritus | 6 mo

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University Hemodialysis Center, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264